CLINICAL TRIAL: NCT01554423
Title: Four-Arm RCT of Brief MI vs. Couples-Based HIV/STI Prevention in South Africa
Brief Title: Four-Arm Randomized Control Trial of Brief MI Versus Couples-Based HIV/STI Prevention in South Africa
Acronym: SA R01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The City College of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dr. William Latimer, Professor and Dean, The City College of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA029894 (NIH); R01DA029894 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-03-15 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: HIV Prevention
Keywords: HIV Prevention Intervention
MeSH Terms: interventions — Counseling; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Testing and Counseling (Active Comparator): One of the four RCT arms will be comprised of couples randomly assigned to testing and counseling on HIV and associated STI co-infections based on revised procedures developed by the CDC. Couples will receive information on the transmission and prevention of HIV and STIs, the meaning of test results, and health consequences. Randomized trial studies of behavioral interventions have incorporated testing and counseling as a comparison condition and studies in the US and SSA countries have shown that testing and counseling on its own can help to reduce HIV/STI risk behaviors.
  Interventions: Other: Testing and Counseling
- Brief Motivational Interview (BMI) (Experimental): The brief motivational interview (BMI) to be tested in the RCT in Pretoria is a one-session, 45 minute intervention that will coordinate three, 15-minute modules with one module each to (1) reduce hazardous drinking; (2) reduce illicit drug use; and (3) promote condom use. Each module is delivered by the clinician using a two-sided laminated card that includes scripted questions and visual aids. Consistent with brief intervention models, the BMI intervention is delivered during one 45 minute session with advice giving as a primary characteristic. Motivational interviewing is also incorporated within the BMI intervention by using a client-centered method of communication to foster behavior change through five techniques of expressing empathy, developing discrepancy, avoiding argumentation, supporting self-efficacy, and motivational rules.
  Interventions: Behavioral: Brief Motivational Interview (BMI)
- Integrated Family and Cognitive Behavioral Therapy (Experimental): The IFCBT model is 6 sessions in length and coordinates the delivery of 4 cognitive-behavioral group couples' sessions with 2 individual couples' sessions to prevent HIV and STI co-infections among adult drug users. IFCBT targets HIV risk and protective factors that operate across multiple ecological systems. The four group couples' sessions coordinate Rational Emotive Therapy and Problem Solving Therapy strategies to reduce HIV risk behavior and promote protective behaviors. The two individual couples' sessions utilize structural and strategic approaches to promote adaptive communication and shared responsibility for condom use and gender equality and to directly address and reduce any form of abuse between partners when present. The six IFCBT sessions are delivered during a 2-week period with two group couples' sessions and one individual couples' session each week.
  Interventions: Behavioral: Integrated Family and Cognitive Behavioral Therapy
- BMI + IFCBT (Experimental): Participants assigned to this experimental arm will receive Brief Motivational Interviewing combined with Integrated Family and Cognitive Behavioral Therapy.
  Interventions: Behavioral: Brief Motivational Interview (BMI); Behavioral: Integrated Family and Cognitive Behavioral Therapy

INTERVENTIONS:
Other: Testing and Counseling — Couples will receive information on the transmission and prevention of HIV and STIs, the meaning of test results, and health consequences.
  Arms: Testing and Counseling
Behavioral: Brief Motivational Interview (BMI) — The brief motivational interview (BMI) to be tested in the RCT in Pretoria is a one-session, 45 minute intervention that will coordinate three, 15-minute modules with one module each to (1) reduce hazardous drinking; (2) reduce illicit drug use; and (3) promote condom use.
  Arms: BMI + IFCBT; Brief Motivational Interview (BMI)
Behavioral: Integrated Family and Cognitive Behavioral Therapy — The IFCBT model is 6 sessions in length and coordinates the delivery of 4 cognitive-behavioral group couples' sessions with 2 individual couples' sessions to prevent HIV and STI co-infections among adult drug users. IFCBT targets HIV risk and protective factors that operate across multiple ecological systems. The four group couples' sessions coordinate Rational Emotive Therapy and Problem Solving Therapy strategies to reduce HIV risk behavior and promote protective behaviors. The two individual couples' sessions utilize structural and strategic approaches to promote adaptive communication and shared responsibility for condom use and gender equality and to directly address and reduce any form of abuse between partners when present.
  Arms: BMI + IFCBT; Integrated Family and Cognitive Behavioral Therapy

SUMMARY:
This study is a Randomized Controlled Trial (RCT) of Integrated and Cognitive Behavioral Therapy for HIV Prevention in Pretoria, South Africa. The RCT will evaluate the efficacy of a brief motivational interview (BMI) and a cognitive-behavioral couples' (IFCBT) intervention alone and in combination against a comparison condition to reduce new cases of HIV and sexually transmitted infections and increase condom use and decrease sexual risk behavior, drug use, and intimate partner violence among young female drug users in Pretoria, South Africa and their primary intimate partners. In the RCT, 384 couples comprised of young female drug users who do (N = 192) and do not (N = 192) trade sex and their primary intimate heterosexual partners will be randomly assigned to one-of-four conditions: (1) testing and counseling; (2) brief motivational interview (BMI); (3) cognitive-behavioral couples' intervention (IFCBT); or (4) BMI and IFCBT combined. Eligibility criteria for couples include an HIV-negative drug using female aged 18 to 40 and their primary intimate partner or spouse who is also HIV negative. Each partner of each couple will be administered assessments with a rapid test for HIV and urine tests for Chlamydia, gonorrhea, trichomoniasis, and drug use at baseline and 3-month, 6-month, and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Live in the Pretoria, South Africa region
* 18-40 Years of Age
* In a steady, intimate relationship for 6 months or longer
* Used illicit drugs in the past 6 months

Exclusion Criteria:

* Acute suicidality/homicidality

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 464 (Actual)
Dates: Start 2010-07; Primary Completion 2017-01-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Biologically confirmed infectious disease status | Outcome measure will be assessed up to 18 months after enrollment.
  Biologically confirmed infectious disease (HIV, Chlamydia, gonorrhea, and trichomoniasis)
Condom use and sexual risk behavior | Outcome measure will be assessed up to 18 months after enrollment.
  Condom use during last sexual intercourse, proportion of unprotected sex episodes; number of partners.
Drug taking risk behavior | Outcome measure will be assessed up to 18 months after enrollment.
  Hazardous alcohol use, and positive urinalysis for marijuana, cocaine, heroin.
Intimate partner violence | Outcome measure will be assessed up to 18 months after enrollment.
  Psychological, physical, and sexual violence.

CONTACTS AND LOCATIONS:
Overall Officials: William W Latimer, Ph.D., Study Director — University of Florida
Locations (1):
- Louis Pasteur Medical Centre, Pretoria, Gauteng, South Africa